CLINICAL TRIAL: NCT00536003
Title: Prevention of Preterm Delivery With Vaginal Progesterone in Women With Preterm Labor
Brief Title: Vaginal Progesterone to Prevent Preterm Delivery in Women With Preterm Labor
Acronym: 4P
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: begoña Martinez de Tejada (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other); Insel Gruppe AG, University Hospital Bern (Other); Basel Women's University Hospital (Other); University of Zurich (Other); Kantonsspital Graubuenden (Other); Cantonal Hospital of St. Gallen (Other); Luzerner Kantonsspital (Other); Kantonsspital Winterthur KSW (Other); Besins Laboratory, Belgium (Unknown); Hospital Bernardino Rivadavia Buenos Aires (Unknown); Hospital Carlos G. Durand Buenos Aires (Unknown); CEMIC Buenos Aires (Unknown); Hospital Donación Francisco Santojanni (Other); Hospital General de Agudos "Dr. Cosme Argerich" (Other); Hospital Dr. T. Alvarez Buenos Aires (Unknown); Hospital Italiano de Buenos Aires (Other); Hospital General de Agudos J. M. Penna (Other); Hospital Materno Infantil Ramón Sardá (Network); Hospital Interzonal Alberto Antranik Eurnekian, provincia Buenos Aires (Unknown); Hospital Municipal Materno Infantil Comodoro Hugo Cesar Meisner, provincia Buenos Aires (Unknown); Hospital Comunal de Tigre, provincia Buenos Aires (Unknown); Hospital Dr. Arturo Oñativia, provincia Buenos Aires (Unknown); Hospital Dr. Carlos Bocalandro, provincia Buenos Aires (Unknown); Hospital Héroes de Malvinas, provincia Buenos Aires (Unknown); Hospital Provincial Magdalena V. de Martínez (Other); Hospital Mariano y Luciano de la Vega, provincia Buenos Aires (Unknown); Hospital Municipal Ostaciana B. de Lavignolle, provincia Buenos Aires (Unknown); Hospital Materno Infantil de San Isidro, provincia Buenos Aires (Unknown); Hospital Virgen del Carmen, provincia Buenos Aires (Unknown); Hospital J. B. Iturraspe, Santa Fe (Unknown); Hospital Maternidad Nuestra Señora De Las Mercedes, Tucumán (Unknown); Hospital Materno Infantil San Roque, Entre Ríos (Unknown); Hospital Villa Dolores, Córdoba (Unknown)
Responsible Party: Sponsor-Investigator, begoña Martinez de Tejada, MD, PhD, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CER: 04-196; matped 04-001
Record Dates: First submitted 2007-09-24; First posted 2007-09-27 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Preterm Delivery; Morbidity; Perinatal Mortality
Keywords: preterm delivery; preterm labor; perinatal morbidity; perinatal mortality
MeSH Terms: conditions — Premature Birth; Perinatal Death; Obstetric Labor, Premature | interventions — Progesterone; Utrogestan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: progesterone
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: progesterone — vaginal capsules containing 200 mg of natural progesterone, once a day, until 36 6/7 weeks of gestation or until preterm delivery (whichever occurs first).
  Other Names: Utrogestan
  Arms: 1
Drug: placebo — vaginal capsules containing placebo, once a day, until 36 6/7 weeks of gestation or until preterm delivery (whichever occurs first).
  Arms: 2

SUMMARY:
The administration of vaginal progesterone, in addition to standard tocolysis, will decrease the risk of delivering prematurely and of recurrent preterm labor. We also hypothesize that the reduction in preterm delivery will be associated with a decrease in infant mortality and morbidity.

DETAILED DESCRIPTION:
The principal aim is to demonstrate that progesterone reduces preterm birth before 37 weeks of gestation. Secondary aims are to show that progesterone 1) reduces preterm birth before 32 and before 34 weeks of gestation 2) reduces the number and duration of recurring episodes of preterm labor and 3) reduces infant mortality and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 240/7 et 336/7 weeks of gestation (based on a reliable estimate by ultrasound performed before 22 weeks)
* Singleton pregnancy
* Intact membranes
* Preterm labor defined as:

  * 2 or more regular and painful uterine contractions in 10 minutes plus one or plus of the following criteria:
  * short cervix detected by vaginal ultrasound scanning (cervical length less than 30 mm until 31 weeks and less than 25 mm from 32 weeks)
  * cervical changes detected clinically (cervical length less or equal 10 mm or Bishop score less than 6
  * cervical changes during hospitalization (more or equal 5 mm between two clinical or US exams)
  * positive fetal fibronectin
* Age ≥ 18 years old
* Signed informed consent
* Possible and accepted follow-up

Exclusion Criteria:

* Multiple gestation
* Cervical cerclage
* Hydramnios (AFI >95th percentile for gestational age or greatest pocket >8 cm)
* Premature rupture of membranes
* Chorioamnionitis (criteria for clinical diagnosis are: elevated WBC, elevated CRP, maternal tachycardia, fetal tachycardia, uterine tenderness and/or amniotic fluid foul odor)
* Cervical dilatation > 3 cm
* Placenta praevia or abruptio placentae
* Intra-uterine growth restriction or non-reassuring fetal status
* Pre-eclampsia or severe hypertension
* Any other maternal or fetal pathology which should indicate medically preterm delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2006-07; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The principal aim is to demonstrate that progesterone reduces preterm birth before 37 weeks of gestation | end of pregnancy

SECONDARY OUTCOMES:
Secondary aims are to show that progesterone 1) reduces preterm birth before 32 and before 34 weeks of gestation 2) reduces the number and duration of recurring episodes of preterm labor and 3) reduces perinatal mortality and morbidity, 4)Side effects | end of pregnancy and 28 days after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Begona Martinez de Tejada, MD, PhD, Principal Investigator — University Hospital, Geneva
Locations (33):
- Argentina (24):
  - Hospital Interzonal Alberto Antranik Eurnekian, Buenos Aires, Alem 349, Ezeiza, Provincia de Buenos Aires
  - Hospital Carlos G. Durand, Buenos Aires, Av. Diaz Velez 5044, Cuidad Autónoma de Buenos Aires
  - Instituto Universitario CEMIC, Buenos Aires, Av. E. Galván 4102, Ciudad Autónoma de Buenos Aires
  - Hospital Bernardino Rivadavia, Buenos Aires, Av. Las Heras 2670, Cuidad Autónoma de Buenos Aires
  - Hospital Mariano y Luciano de la Vega, Buenos Aires, Av. Libertador 710, Moreno, Provincia de Buenos Aires
  - Hospital Maternidad Nuestra Señora De Las Mercedes, Buenos Aires, Av. Mate de Luna 1555, Provincia de Tucumán
  - Hospital Villa Dolores, Buenos Aires, Belgrano 1500, Villa Dolores, Provincia de Códoba
  - Hospital J. B. Iturraspe, Buenos Aires, Bvd. Pellegrini 3551, Provincia de Santa Fe
  - Hospital Comunal de Tigre, Buenos Aires, Casareto 118, Tigre, Provincia de Buenos Aires
  - Hospital Materno Infantil de San Isidro, Buenos Aires, Diego Palma 505, San Isidro, Provincia de Buenos Aires
  - Hospital Virgen del Carmen, Buenos Aires, Dr. Félix Pagola 1502, Zárate, Provincia de Buenos Aires
  - Hospital Dr. T. Alvarez, Buenos Aires, Dr. Juan Felipe Aranguren 2701, Cuidad Autónoma de B.A.
  - Hospital Materno Infantil Ramón Sardá, Buenos Aires, Esteban de Luca 2151, Ciudad Autónoma de Buenos Aires
  - Hospital Municipal Materno Infantil Comodoro Meisner, Buenos Aires, Iparaguirre Nº 239, Pte. Derqui, Provincia de Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires, Juan D. Perón 4190, Ciudad Autónoma de Buenos Aires
  - Hospital Materno Infantil San Roque, Buenos Aires, La Paz 435, Provincia de Entre Ríos
  - Hospital Municipal Ostaciana B. de Lavignolle, Buenos Aires, Monte 848, Morón, Provincia de Buenos Aires
  - Hospital J. M. Penna, Buenos Aires, Pedro Chutro 3380, Cuidad Autónoma de Buenos Aires
  - Hospital Donación Francisco Santojanni, Buenos Aires, Pilar 950, Ciudad Autónoma de Buenos Aires
  - Hospital Dr. Cosme Argerich, Buenos Aires, Py Y Margall 750, Cuidad Autónoma de Buenos Aires
  - Hospital Dr. Arturo Oñativia, Buenos Aires, Ramón Carillo 1339, Rafael Calzada, Provincia de Buenos Aires
  - Hospital Héroes de Malvinas, Buenos Aires, Ricardo Balbín 1910, Merlo, Provincia de Buenos Aires
  - Hospital Magdalena V. de Martínez, Buenos Aires, Rura 9 Constituyentes 395, Gral, Pacheco, Provincia de B.A.
  - Hospital Dr. Carlos Bocalandro, Buenos Aires, Ruta 8Km. 20,5 N°9100, Loma Hermosa, Provincia de Buenos Aires
- Switzerland (9):
  - Universitäts-Frauenklinik Kantonespital Basel, Basel, Basel
  - Universitätsfrauenklinik Bern, Bern, Canton of Bern
  - Maternity of the University Hospital of Geneva, Geneva, Canton of Geneva
  - Frauenklinik Kantonspital Luzern, Lucerne, Canton of Lucerne
  - Frauenklinik Kantonspital St Gallen, Sankt Gallen, Canton of St. Gallen
  - University Hospital Zürich, Zurich, Canton of Zurich
  - Kantonales Frauenspital Chur, Chur, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne, Lausanne
  - Frauenklinik Kantonspital Winterthur, Winterthur, Winterthur

REFERENCES:
- [Derived] Martinez de Tejada B, Karolinski A, Ocampo MC, Laterra C, Hosli I, Fernandez D, Surbek D, Huespe M, Drack G, Bunader A, Rouillier S, Lopez de Degani G, Seidenstein E, Prentl E, Anton J, Krahenmann F, Nowacki D, Poncelas M, Nassif JC, Papera R, Tuma C, Espoile R, Tiberio O, Breccia G, Messina A, Peker B, Schinner E, Mol BW, Kanterewicz L, Wainer V, Boulvain M, Othenin-Girard V, Bertolino MV, Irion O; 4P trial group. Prevention of preterm delivery with vaginal progesterone in women with preterm labour (4P): randomised double-blind placebo-controlled trial. BJOG. 2015 Jan;122(1):80-91. doi: 10.1111/1471-0528.13061. Epub 2014 Sep 11. PMID 25209926